CLINICAL TRIAL: NCT01508663
Title: The Beneficial Role of Percutaneous Coronary Intervention Over Optimal Medical Therapy in Elderly Patients (Age > 75 Years Old) With Coronary Artery Disease: a Randomized Controlled Study
Brief Title: The Beneficial Role of Percutaneous Coronary Intervention Over Optimal Medical Therapy in Elderly Patients With Coronary Artery Disease
Acronym: BRAVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Myeong-Ki Hong, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2010-0016
Record Dates: First submitted 2012-01-03; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease 75years of age or older
MeSH Terms: conditions — Coronary Artery Disease | interventions — Calcium Channel Blockers; Angiotensin-Converting Enzyme Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Nitrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI+OMT group (Experimental): PCI (Everolimus Eluting Stent or Zotalolimus Eluting Stent) added to OMT after randomization and follow up for 12 months
  Interventions: Device: Everolimus Eluting Stent or Zotalolimus Eluting Stent
- OMT alone group (Active Comparator): OMT alone after randomization and follow up for 12 months
  Interventions: Drug: ARB, CCB, ACE-inhibitor, statin, Nitrate, Antiplate etc.

INTERVENTIONS:
Device: Everolimus Eluting Stent or Zotalolimus Eluting Stent — Everolimus Eluting Stent(Xience V, Xience prime) Zotalolimus Eluting Stent(Endeavor-resolute, Resolute Integrity)
  Arms: PCI+OMT group
Drug: ARB, CCB, ACE-inhibitor, statin, Nitrate, Antiplate etc. — one or two anti-platelet agents, beta-blockers, calcium channel blockers, nitrates, angiotensin converting enzyme inhibitors (ACEIs) or angiotensin receptor blockers (ARBs), and statin
  Arms: OMT alone group

SUMMARY:
The primary purpose of this study is to determine whether PCI added to OMT could be superior over OMT alone in the prevention of late adverse cardiac and cerebro-vascular events in elderly patients with coronary artery disease (CAD) during the additional 12 months.

DETAILED DESCRIPTION:
Study Design

* Prospective, randomized, multi-center study of each 1600 subjects enrolled.
* Eligible subjects will be randomized 1:1 to a) PCI added to OMT (n=800) vs. b) OMT alone(n=800).

Subsequently, subjects in PCI added to OMT group will be randomly assigned to everolimus eluting stent(n=400) vs. zotarolimus eluting sten(n=400). All subjects will be followed for 1 year after randomization. Additional long-term follow-up (2- or 3-year) will be preceded in the next plan after 1-year study period.

* Subjects with CAD who meet all inclusion and exclusion criteria will be included
* Clinical and laboratory follow-up should be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CAD and those in whom initial CCS class I to III angina or Braunwald classification less than IIB
2. Patients with age 75 years or older
3. Patients receiving OMT (one or two anti-platelet agents, beta-blockers, calcium channel blockers, nitrates, angiotensin converting enzyme inhibitors (ACEIs) or angiotensin receptor blockers (ARBs), and statin)
4. Patients with stenosis of at least 70% in at least one proximal epicardial coronary artery or objective evidence of myocardial ischemia (substantial changes in ST-segment depression or T-wave inversion on the resting electrocardiogram or inducible ischemia with either exercise or pharmacologic vasodilator stress)
5. Patients with signed informed consent

Exclusion Criteria:

1. Patients with persistence of CCS IV angina
2. Resting chest pain (≥ Braunwald classification IIB)
3. Patients who experienced a markedly positive stress test (substantial ST- segment depression or hypotensive response during stage 1 of the Bruce protocol)
4. Patients with age 85 years or older
5. Patients with refractory CHF or cardiogenic shock
6. Patients with an EF of less than 30%
7. Patients who have received revascularization within the previous 6 months
8. Patients with coronary anatomy not suitable for PCI
9. Life expectancy ≤ 2 year

Ages: 75 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event | 12month
  The primary end-point is the occurrence of major adverse cardiac event [cardiovascular death, non-fatal MI (excluding periprocedural MI), stroke or any revascularization (PCI or coronary bypass surgery [CABG]) for 12 months following the randomization to the assigned management]

SECONDARY OUTCOMES:
cardiac or non-cardiac major adverse event | 12month
  1. The composite of cardiac or non-cardiac death, non-fatal MI, stent thrombosis (ST), target vessel revascularization (TVR) (either by PCI or CABG), non-TVR, hospitalization for unstable angina pectoris (UAP) or congestive heart failure (CHF), and cerebrovascular accident (CVA) for 12 months.
  2. Major determinant for the occurrence of major events
  3. Sub-study according to the subsets of disease
  4. Association between parameters at index procedure and clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Myeong-Ki, Hong, Seoul, South Korea